CLINICAL TRIAL: NCT02313636
Title: Narrow Band Imaging in Flexible Cystocopy - DaBlaCa-7
Brief Title: Narrow Band Imaging in Flexible Cystocopy
Acronym: DaBlaCa-7
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Herlev Hospital (Other); Hospitalsenheden Vest (Other); Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Other Study IDs: DaBlaCa-7
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2023-05-31 (Actual); Status verified 2023-05

CONDITIONS: Narrow Band Imaging in Flexible Cystoscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Patients with first time hematuria or patients previously diagnosed with papillomas/CIS of the bladder are included in the study. All surgeons are highly experienced in WL cystoscopy and familiar with NBI findings. Cystoscopy is performed with HD cameras and Olympus light sources.

First, a systematic cystoscopy is made in WL. Secondly, the clinical decision is noted. After WL, the cystoscopy is made with NBI and any potential subsequent change in the clinical decision is noted.

A total number of 896 patients is planned to be included.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing flexible cystoscopy because of haematuria or previous NMIBC

Exclusion Criteria:

* Patients not fullfilling the above

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing flexible cystoscopy because of haematuria or previous NMIBC
Sampling Method: Non-Probability Sample
Enrollment: 955 (Actual)
Dates: Start 2014-05; Primary Completion 2015-07 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
change in the clinical decision | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Bjerggaard Jensen, DMSc, Principal Investigator — University of Aarhus
Locations (3):
- Denmark (3):
  - Aarhus University Hospital, Århus N
  - Herlev Hospital, Herlev
  - Hospitalsenheden Vest, Holstebro